CLINICAL TRIAL: NCT07220564
Title: Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Multiple Ascending Peroral Doses of Inno8 in People With Haemophilia A
Brief Title: A Research Study Looking at How Different Doses of Study Medicine (Inno8) Work in the Body of People With Haemophilia A
Acronym: VOYAGER2
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NN7442-8454; U1111-1317-4366 (Other: Universal Trial Number); 2025-520490-38 (EudraCT Number)
Record Dates: First submitted 2025-10-22; First posted 2025-10-24 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Haemophilia A
MeSH Terms: conditions — Hemophilia A

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1 (Experimental): Participants will receive oral dose of NNC0442-0344 A.
  Interventions: Drug: NNC0442-0344 A
- Cohort 2 (Experimental): Participants will receive oral dose of NNC0442-0344 A.
  Interventions: Drug: NNC0442-0344 A

INTERVENTIONS:
Drug: NNC0442-0344 A — NNC0442-0344 A will be administered orally.
  Other Names: Inno8

SUMMARY:
This study will test how different doses of study medicine (Inno8) work in the bodies of people with haemophilia A. The purpose of the study is to see if Inno8 is safe to use for people with haemophilia A. The study medicine is a new medicine that cannot yet be prescribed by doctors. The study will last for about 11 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Age 18-64 years (both inclusive) at the time of signing the informed consent.
* Body weight greater than or equal to (≥) 45 kilograms (kgs).
* Diagnosis of congenital haemophilia A with factor VIII (FVIII) activity less than or equal to (≤) 15 percentage (%) with or without FVIII inhibitors, based on medical records.

Exclusion Criteria:

* Current or prior exposure to any prophylactic treatment for haemophilia A within 5 half-lives of the medicinal product by the time of screening.
* Body mass index ≥30.0 kilogram per square meter (kg/m^2).
* Increased risk of thrombosis, e.g. known history of personal or first-degree relative(s) with unprovoked deep vein thrombosis.
* Any clinical signs or established diagnosis of venous or arterial thromboembolic disease.
* Any known coagulation disorders other than haemophilia A.
* Ongoing or planned immune tolerance induction therapy.
* Presence of clinically significant gastrointestinal disorders potentially affecting absorption of drugs and/or nutrients, as judged by the investigator.

Ages: 18 Years to 64 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-10-23 (Actual); Primary Completion 2026-12-21 (Estimated); Study Completion 2026-12-21 (Estimated)

PRIMARY OUTCOMES:
Number of treatment emergent adverse events | From time of dosing (Day 1) to end of follow-up (Day 46)
  Measured as count of events.

SECONDARY OUTCOMES:
Change in D-dimer | From time of dosing (Day 1) to end of follow-up (Day 46)
  Measured as absolute and percentage (%).
Change in prothrombin fragment 1 and 2 | From time of dosing (Day 1) to end of follow-up (Day 46)
  Measured as absolute and %.
Change in fibrinogen | From time of dosing (Day 1) to end of follow-up (Day 46)
  Measured as absolute and %.
Change in platelets | From time of dosing (Day 1) to end of follow-up (Day 46)
  Measured as absolute and %.
Occurrence of anti-Inno8 antibodies | From time of dosing (Day 1) to end of follow-up (Day 46)
  Measured as count.
Cmax: the maximum concentration of Inno8 after multiple doses | From Day 10 to Day 11
  Measured as nanograms per millilitre (ng/mL).
Tmax: the time to Cmax after last multiple dose | From day 10 to Day 11
  Measured as hours.
Tmax: the time to Cmax after first dose | From Day 1 to Day 2
  Measured as hours.
AUC: the area under the Inno8 concentration-time curve in the dosing interval after multiple doses | From Day 10 to Day 11
  Measured as nanograms*day per millilitre (ng*day/mL).
Maximum thrombin generation (peak height) | From Day 10 to Day 11
  Measured as nanomolar (nM).

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 2834), Study Director — Novo Nordisk A/S
Locations (18):
- United States (3):
  - Indiana Hemophilia-Thromb Ctr, Indianapolis, Indiana
  - University of Iowa_Iowa City, Iowa City, Iowa
  - Penn State MS Hershey Med Ctr, Hershey, Pennsylvania
- Austria (2):
  - Universitätsklinik für Innere Medizin V, Innsbruck
  - AKH - Klin. Abt. f. Haematologie u. Haemostaseologie, Vienna
- Germany (2):
  - Vivantes Netzwerk für Gesundheit GmbH - Vivantes Klinikum im Friedrichshain, Berlin
  - Medizinische Hochschule Hannover - Hämatologie, Hämostaseologie, Onkologie, Hanover
- Italy (2):
  - AOU Careggi Firenze, Florence
  - Azienda Ospedaliera Universitaria Federico II di Napoli, Napoli
- Poland (3):
  - Uniwersytecki Szpital Kliniczny w Bialymstoku, Bialystok
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - Instytut Hematologii i Transfuzjologii, Warsaw
- Spain (4):
  - Hospital Vall d'Hebron, Barcelona
  - Hospital Universitario La Paz, Madrid
  - Hospital Regional Universitario de Málaga, Málaga
  - Hospital Clinico Universitario de Salamanca, Salamanca
- United Kingdom (2):
  - West Midlands Adult Comprehensive Care Haemophilia, Birmingham
  - Royal Free Hospital - Haemophilia, London

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: https://novonordisk-trials.com